CLINICAL TRIAL: NCT06100276
Title: A Phase 1/2, Multicenter, Single Ascending Dose Study to Evaluate the Safety, Tolerability, and Exploratory Efficacy of Intrathecally Administered Gene Therapy AMT-162 in Adult Participants With SOD1 Amyotrophic Lateral Sclerosis (SOD1-ALS).
Brief Title: Safety, Tolerability, and Exploratory Efficacy Study of Intrathecally Administered Gene Therapy AMT-162 in Adult Participants With SOD1 Amyotrophic Lateral Sclerosis (SOD1-ALS)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UniQure Biopharma B.V. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AMT-162-001
Record Dates: First submitted 2023-10-20; First posted 2023-10-25 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Gene Therapy; AAV (adeno-associated virus); ALS; SOD1
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3 single Ascending Dose Levels (Experimental): Experimental: 3 single Ascending Dose Levels
  The study will be open-label with an initial plan to explore 3 dose levels of AMT-162 in approximately 6 to 12 Participants in total. Each Participant will receive a single dose of AMT-162 delivered via an intrathecal (IT) infusion and will be followed for up to 5 years after AMT-162 administration.
  Interventions: Drug: AMT-162
- EXPANSION COHORT (Experimental): Expansion cohort: To further test selected dose from the SAD part in approximately 6 to 8 participants
  The study will be open-label. Each Participant will receive a single dose of AMT-162 delivered via an intrathecal (IT) infusion and will be followed for up to 5 years after AMT-162 administration.
  Interventions: Drug: AMT-162

INTERVENTIONS:
Drug: AMT-162 — AMT-162, the investigational product (IP), is a nonreplicating, rep/cap-deleted, self-complementary Recombinant adeno-associated virus (rAAV) vector based on adeno-associated virus (AAV) serotype rh10 and contains complementary deoxyribonucleic acid (cDNA) encoding an artificial miRNA targeting the SOD1 gene.

SUMMARY:
This is the study of AMT-162 in Participants with SOD1-ALS and is designed to evaluate the safety, tolerability, and exploratory efficacy of intrathecally administered gene therapy AMT-162. AMT-162-001 is a Phase 1/2, multi-center, single ascending dose study.

DETAILED DESCRIPTION:
AMT-162 is an investigational gene therapy that encodes an artificial microribonucleic acid (microRNA or miRNA) targeting the SOD1 gene. This clinical study will test the safety of AMT-162 and explore the hypothesis that it will silence expression of mutant cytosolic SOD1 and thereby ameliorate the course of ALS caused by this mutant gene.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed clinical and genetic diagnosis of SOD1-mediated ALS (SOD1-ALS) experiencing signs and/or symptoms of lower motor neuron dysfunction (weakness, atrophy, cramps, fasciculations), with or without upper motor neuron symptoms (weakness, bring reflexes, spasticity).
* ALSFRS-R score ≥ 25 at Screening.
* Slow vital capacity (SVC) ≥50% of predicted normal value.
* Capable of providing informed consent and complying with trial procedures, including: medically able to undergo lumbar puncture and has a responsible caregiver able to attend all clinic visit with the Participant.

Exclusion Criteria:

* SOD1 pathogenic or likely pathogenic variants in amino acid regions 43-47.
* Pathogenic repeat expansion in the C9orf72 gene
* Any of the following prior or concomitant treatments:

  * Any prior SOD1 suppression therapy with viral microRNA mediators
  * Prior SOD suppression therapy with antisense oligonucleotide (ASO) mediators such as tofersen (QALSODY™). Exception: Patients who previously received tofersen may be enrolled if the last dose of tofersen was received at least 20 weeks prior to the first Screening assessment and if there were no previous tofersen-related SAEs or ongoing tofersen-related adverse events that would increase the risk of receiving AMT-162, per Investigator judgment.
  * Other ALS medications riluzole (RILUTEK®, TIGLUTIK®), edaravone (RADICAVA®), and sodium phenylbutyrate and taururosdiol combination (RELYVRIO) or bioequivalents are allowed if dose is stable for 30 days prior to immunosuppression.
  * Any prior administration of an AAV gene therapy.
* Participants must be willing to forego new ALS treatments through at least 6 months after infusion of AMT-162. After 6 months, Investigators and participants may decide to add new ALS medications or change existing ALS medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of ascending doses of intrathecally administered AMT-162 in Participants with SOD1-ALS | up to 5 years
  Occurrence of TEAEs upon administration of ascending doses of AMT-162

SECONDARY OUTCOMES:
Characterization of Immune Response to AMT-162 and Shedding of intrathecally administered AMT-162. | up to 5 years
  Any positive results in shedding samples will be summarized at each timepoint. Immunogenicity parameters will be summarized for each visit.
Characterization of the Effect of intrathecally administered AMT-162 | up to 5 years
  Change from Baseline in Slow Vital Capacity (SVC) percent of predict value, Hand-held dynamometry (HHD) scores, and Neurofilament light chain (NfL) protein levels in serum.
  Immunogenicity parameters will be summarized for each visit.

CONTACTS AND LOCATIONS:
Overall Officials: Executive Director, Clinical Development, Study Director — UniQure Biopharma B.V.
Locations (12):
- United States (11):
  - Barrow Neurological Institute, Phoenix, Arizona
  - University of California Irvine, Irvine, California
  - California Pacific Medical Center, San Francisco, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - University of Kansas Medical Center, Fairway, Kansas
  - Massachusetts General Hospital, Sean M. Healey and AMG Center for ALS Research, Boston, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Columbia University Irving Medical Center, New York, New York
  - University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania
- Norrlands Universitetssjukhus, Umeå, Vasterbottens Ian, Sweden

IPD SHARING:
Plan to Share IPD: No